CLINICAL TRIAL: NCT06393478
Title: Southeastern Europe Microcirculation Registry
Acronym: SATURATION
Status: Recruiting | Type: Observational
Sponsor: Institute for Cardiovascular Diseases Dedinje (Other)
Collaborators: Abbott Medical Devices (Industry)
Responsible Party: Principal Investigator, Ivan Ilić, MD, PhD, Assistant Professor, Institute for Cardiovascular Diseases Dedinje
Other Study IDs: IKVBD-KARD-001
Record Dates: First submitted 2024-04-26; First posted 2024-05-01 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Angina, Microvascular; Coronary Microvascular Dysfunction; Coronary Artery Disease
Keywords: microvascular angina, thermodilution, coronary flow reserve
MeSH Terms: conditions — Microvascular Angina; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
SATURATION is a prospective multicenter registry of consecutive patients who undergo coronary physiology testing using Pressure Wire X and Coroflow Coroventis Cardiovascular System software (Abbott Vascular, Abbott Park, IL, USA) and to assess the regional practice of patient selection, cardiovascular outcomes and additional procedures (stress testing, angiography, etc.) done after comprehensive invasive coronary physiology evaluation.

DETAILED DESCRIPTION:
The study will include adults of both sexes older than 18 years with angina symptoms or angina equivalent referred to cath lab for evaluation of coronary artery disease (CAD) that underwent invasive physiology testing performed (microcirculation testing +/- vasospasm testing) using Coroflow Coroventis Cardiovascular system (Abbott Vascular, Abbott Park, IL, USA) The study will exclude persons under the age of 18, pregnant of nursing ant the ones where no coronary physiology measurements performed

.

The following data will be collected at enrollment:

* De-identified demographic data
* Cardiovascular risk factors and significant co-morbidities
* Laboratory investigations of interest
* Prior cardiovascular events
* Pre-procedure medications
* Echocardiogram within 3 months of invasive coronary procedure
* Non-invasive ischemia testing within 3 months of invasive coronary procedure
* Seattle Angina Questionnaire (SAQ)
* EQ-5D-5L
* Details of the coronary angiography and invasive physiology procedure including procedural complications
* Post-procedure medications

Data that will be collected during invasive coronary physiology testing:

Vasospastic angina testing (which artery, what test, result) Microvascular angina testing (which artery, CFR, IMR, RRR, FFR, Pd, Pa and all transit times)

Patients will be seen at follow up visits and the following data will be collected every 6 months for up to 5 years:

* Major adverse cardiovascular events including repeat invasive coronary angiography since last follow up
* Current medications
* SAQ
* EQ-5D-5L
* Non-invasive ischemia testing since last follow up Outcomes will be evaluated every 6 months for 5 years via direct patient contact by research staff or at follow up visits. Outcomes will be collected based on existing medical documentation.

Primary outcomes:

* all-cause death and non-fatal MI
* composite MACE: all-cause death, non-fatal MI, coronary revascularization, hospitalization for cardiovascular causes (acute coronary syndrome, heart failure, angina, repeated coronary angiography) Secondary outcomes: all-cause death, cardiovascular death, MI, coronary revascularization, stroke, hospitalization for heart failure, hospitalization for acute coronary syndrome, repeated coronary angiography

Patient-centered outcomes:

* Freedom from angina (SAQ questionnaire)
* Quality of life using EQ-5D-5L questionnaire
* Follow up non-invasive ischemia testing (if performed)

ELIGIBILITY:
Inclusion Criteria:

* Adults of both sexes older than 18 years
* Angina symptoms or angina equivalent
* Referred to Cath lab for evaluation of CAD
* Invasive physiology testing performed (microcirculation testing +/- vasospasm testing) using Coroflow Coroventis Cardiovascular system (Abbott Vascular, Abbott Park, IL, USA)

Exclusion Criteria:

* Persons under the age of 18
* Pregnant of nursing
* No coronary physiology measurements performed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients suffering from angina who undergo coronary physiology testing using Pressure Wire X and Coroflow Coroventis Cardiovascular System software (Abbott Vascular, Abbott Park, IL, USA).
Sampling Method: Non-Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2029-03-01 (Estimated); Study Completion 2034-03-01 (Estimated)

PRIMARY OUTCOMES:
all-cause death and non-fatal MI | 5 years
  The study will record aggregate number of participants that died and/or suffered from myocardial infarction after invasive physiology procedure
composite MACE | 5 years
  The study will record aggregate number of participants that died from any cause and/or experienced non-fatal myocardial infarction and/or coronary angioplasty procedure and/or hospitalization for cardiovascular causes (acute coronary syndrome, heart failure, angina, repeated coronary angiography)

SECONDARY OUTCOMES:
all-cause death | 5 years
  The study will record number of participants that died after invasive coronary physiology
cardiovascular death | 5 years
  The study will record number of participants that died due to cardiovascular causes after invasive coronary physiology
myocardial infarction | 5 years
  The study will record the number of participants that suffered from myocardial infarction after invasive coronary physiology
coronary revascularization | 5 years
  The study will record number of participants that undergo surgical and/or percutaneous revascularization after invasive coronary physiology
stroke | 5 years
  The study will record the number of participants that suffered from stroke after invasive coronary physiology
hospitalization for heart failure | 5 years
  The study will record the number of participants that are hospitalized for heart failure after invasive coronary physiology
hospitalization for acute coronary syndrome | 5 years
  The study will record the number of participants that are hospitalized for acute coronary syndrome after invasive coronary physiology
repeated coronary angiography | 5 years
  The study will record the number of participants that undergo repeated coronary angiography after invasive coronary physiology

CONTACTS AND LOCATIONS:
Locations (10):
- Croatia (2):
  - CHC Rijeka, Rijeka
  - KBC Zagreb, Zagreb
- Greece (4):
  - MITERA General Hospital, Athens
  - Hippokration Hospital, Athens
  - Heraklion University Hospital, Heraklion
  - University Hospital of Patras, Pátrai
- Tel Aviv Sourasky MC, Tel Aviv, Israel
- Serbia (2):
  - Institute for cardiovascular diseases Dedinje, Belgrade
  - Institute for cardiovascular diseases Vojvodine, Novi Sad
- UMC Ljubljana, Ljubljana, Slovenia

DOCUMENTS (1):
  • Study Protocol (2024-03-21): https://cdn.clinicaltrials.gov/large-docs/78/NCT06393478/Prot_000.pdf